CLINICAL TRIAL: NCT01152684
Title: Complementary & Alternative Care Behavior in HIV+ Latinos in the US-Mexico Border
Brief Title: Complementary & Alternative Medicine Use in HIV+ Latinos in the US-Mexico Border
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: R21AT004676-01A1 (NIH); R21AT004676-01A1 (NIH)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: HIV Positive
Keywords: CAM; HIV-Positive; Latinos; US-Mexico Border region; San Diego-Tijuana; Identify the nature and extent of complementary and alternative medicine use among HIV-positive Latinos in the US-Mexico border region
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV-Positive Latinos living in San Diego or Tijuana: This is an exploratory study of Latinos living with HIV in the San Diego-Tijuana US-Mexico border region.

SUMMARY:
The goal of The investigators community-based participatory research study is to identify the nature and extent of complementary and alternative medicine (CAM) use among HIV-positive Latinos on the San Diego/Tijuana border. CAM use among US Latinos living with HIV is associated with delayed utilization of and poor adherence to antiretroviral therapies (ARVs) that may exacerbate health disparities in HIV care access and health outcomes. This study will lead to development of culturally-effective interventions to improve access and adherence to HIV care in Latinos who face health disparities. The investigators hypothesis is that greater use of CAM will be observed among HIV-positive Latinos who report a) crossing the U.S. border more frequently, and b) having migrated to Tijuana or San Diego (e.g. from southern Mexico). The investigators also hypothesize that compared to HIV-positive Latinos who report using herbal CAM, those who do not use herbal CAM are more likely to be receiving ARVs and report higher levels of adherence to ARVs; Compared to HIV-positive Latinos who do not attend religious services regularly, those who attend religious services regularly are more likely to be receiving ARV; Compared to HIV- positive Latinos who report experiencing HIV related stigma, those who do not report experiencing HIV-related stigma are significantly more likely to be receiving ARVs.

DETAILED DESCRIPTION:
The goal of our community-based participatory research study is to identify the nature and extent of complementary and alternative medicine (CAM) use among HIV-positive Latinos on the San Diego/Tijuana border. CAM utilization among US Latinos living with HIV is associated with delayed utilization of and poor adherence to antiretroviral therapies (ARVs) that may exacerbate health disparities in HIV care access and health outcomes. US Latinos face more barriers to HIV care than non-Latino Whites including less health insurance, delays in seeking HIV care, and entering care at advanced stages of HIV disease. Latinos living with HIV/AIDS may be more likely to use CAM when faced with barriers to accessing conventional HIV care than non-Latino Whites. CAM use, including herbal therapies, seeking care from alternative healers, and religious practices may be implicated in HIV-related health disparities for US Latinos living with HIV, but research is lacking, particularly in the context of binational healthcare utilization. The United States (US)-Mexico border is a demographically booming region characterized by a shared population living on either side of the border and who cross frequently to Tijuana or to San Diego; US HIV care providers working in the USMexico border region serve many Latinos who access services and care on both sides of the border.Concern over clinician reaction to CAM may erode Latino patient-provider communication, yet assessment of CAM use from patient and clinician perspective and health system characteristics is also lacking. We will describe CAM use in HIV-positive Latinos in the US-Mexico border region to improve culturally-effective care delivery and inform future biomedical and behavioral interventions to decrease disparities in ARV access and utilization, and improve HIV-related health outcomes for US Latinos.

Specific aims of our study are:

Aim 1: To assess CAM-specific health care behavior, including bi-national CAM utilization from allied/alternative health personnel (e.g. pharmacists, non-Western medicine healers) among HIV-positive Latinos residing in Tijuana and San Diego.

Hypothesis 1 (H1) Greater use of CAM will be observed among HIV-positive Latinos who report a) crossing the U.S. border more frequently, and b) having migrated to Tijuana or San Diego (e.g. from southern Mexico).

Aim 2: To assess use of CAM in the context of HIV treatment utilization and practices, including factors related to delayed entry into HIV care (e.g. HIV stigma); and access to, utilization of and adherence to ARVs among HIV-positive Latinos residing in Tijuana or San Diego. H2.a) Compared to HIV-positive Latinos who report using herbal CAM, those who do not use herbal CAM are more likely to be using ARVs and report higher levels of adherence to ARVs; H2.b) Compared to HIV-positive Latinos who do not attend religious services regularly, those who attend religious services regularly are more likely to use ARV.

H2.c) Compared to HIV-positive Latinos who report experiencing HIV-related stigma, those who do not report experiencing HIV-related stigma are significantly more likely to use ARVs and report lesser utilization of CAM.

Aim 3: To determine perceived barriers to communicating use of CAM and ARV adherence to clinicians among HIV-positive Latinos residing in Tijuana or San Diego, including satisfaction with clinician communication; concern about physician response to reporting CAM modalities such as herbal therapies, pharmacy practices in Mexico and folk healing perception of ARV efficacy, and perception of ARV efficacy.

H3) Among HIV-positive CAM users, disclosure of CAM use will be higher in Latino patients who report higher satisfaction with communication with clinicians than those who report lower satisfaction with clinicians.

Aim 4: To explore provider and system barriers to culturally-effective communication about CAM and ARV adherence with HIV-positive Latino patients, including clinician knowledge about patient CAM practices.

To address Aims 1-3 we will conduct a quantitative study using interviewer-administered surveys with 200 HIV positive Latinos (100 from each side of the border). In Aim 4 we will purposively sample 20 HIV clinicians on both sides of the border and conduct in-depth interviews. Our aims are consistent with the Office of AIDS Research 2008 Plan to assess sociocultural and structural determinants and health systems that enhance, sustain and/or perpetuate health disparities.7 Capitalizing on our HIV research expertise with Latino communities, this study will lead to development of culturally-effective interventions to improve timeliness and adherence to HIV care in populations with documented health disparities and will reduce gaps in care.

ELIGIBILITY:
Inclusion Criteria:

* Latino
* Speak English or Spanish or both
* Lived in San Diego or Tijuana for at least 1 month in the last year
* 18 years or older
* HIV-positive or living with AIDS

Exclusion Criteria:

* Non-Latino
* Speak neither English nor Spanish
* Have not lived in San Diego or Tijuana for at least 1 month in the last year
* Under 18 years of age
* Not HIV-positive or living with AIDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will be selected from 2 locations: 1. San Diego: San Ysidro Health Center(SYHC) will serve as the recruitment site on the US side of the border. Latinos comprise >90% of SYHC's patient population. SYHC provides HIV primary medical care to over 400 HIV-positive individuals. SYHC's HIV-positive Latino patient population includes persons who may or may not be on ARVs and who participate in clinic services to varying degrees. Previous studies with HIV-positive patients at SYHC indicate cross-border mobility and bi-national care seeking behavior in this clinic population. 2.Tijuana: The Agencia Familiar Binacional (AFABI;Binational Health Agency) opened the first HIV medical and social services agency clinic in Tijuana. This clinic is in close proximity to the municipal health clinic, where a large number of HIV-positive cases are diagnosed, and is linked with other non-profit social services agencies for HIV-positive persons, many of whom face barriers to ARVs.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Zúñiga, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- San Ysidro Health Center, San Ysidro, California, United States